CLINICAL TRIAL: NCT05272709
Title: CURATE: A Cancer Research UK Phase I/II, Dose Escalation and Expansion Trial of TT-702, A Selective Adenosine A2BR Antagonist, Given Orally as a Monotherapy Agent and in Combination, in Patients With Advanced Solid Tumours
Brief Title: TT-702 in Patients With Advanced Solid Tumours.
Acronym: CURATE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Teon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/21/005; 2021-001062-37 (EudraCT Number)
Record Dates: First submitted 2022-02-09; First posted 2022-03-09 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors
Keywords: Adenosine receptors; MSI Deficient Cancers; MMR Deficient Cancer; Castrate resistant Prostate Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1M (Monotherapy escalation cohort) (Experimental): This cohort will recruit patients with solid tumours.
  Interventions: Drug: TT-702
- Cohort 2M: mCRPC (Monotherapy expansion cohort) (Experimental): This cohort will recruit patients with mCRPC only.
  Interventions: Drug: TT-702
- Cohort 2M: MSI/MMR defective tumours (Monotherapy expansion cohort) (Experimental): This cohort will recruit patients with MSI/MMR defective tumours only.
  Interventions: Drug: TT-702
- Cohort 2M: TNBC (Monotherapy expansion cohort) (Experimental): This cohort will recruit patients with TNBC only.
  Interventions: Drug: TT-702
- Cohort 1A (TT-702 + Darolutamide combination escalation cohort) (Experimental): This cohort will recruit patients with mCRPC only.
  Interventions: Drug: TT-702; Drug: Darolutamide
- Cohort 2A (TT-702 + Darolutamide combination expansion cohort) (Experimental): This cohort will recruit patients with mCRPC only.
  Interventions: Drug: TT-702; Drug: Darolutamide

INTERVENTIONS:
Drug: TT-702 — TT-702 will be administered orally, once daily, for up to 12 months.
Drug: Darolutamide — Darolutamide will be administered orally, twice daily, for up to 12 months.
  Arms: Cohort 1A (TT-702 + Darolutamide combination escalation cohort); Cohort 2A (TT-702 + Darolutamide combination expansion cohort)

SUMMARY:
This clinical trial is evaluating the drug candidate TT-702 in patients with advanced solid tumours. The main aims of the trial are to determine the maximum dose of TT-702 that can be given safely to patients alone and in combination with other anti-cancer agents.

DETAILED DESCRIPTION:
TT-702 is a 'small molecule prodrug'. TT-702 is converted into TT-478, which then targets and blocks the function of the 'A2B adenosine receptor'. It is hoped that by blocking this receptor the immune system will become more active in recognising and removing tumour cells.

This clinical trial has two phases:

* Phase I, dose escalation phase - groups of patients will receive increasing doses of TT-702 to find an optimal dose that best targets the tumours. This phase will consist of both monotherapy and combination escalation cohorts. In the combination escalation cohorts, TT-702 will be evaluated in combination with the androgen receptor (AR) antagonist darolutamide to be assessed in mCRPC. Potential agents for further combination escalation cohorts have not yet been defined.
* Phase II, expansion phase - larger groups of patients will receive the selected dose of TT-702 considered to be optimal in the Phase I, dose escalation phase. This phase will consist of three monotherapy expansion cohorts (metastatic castrate resistant prostate cancer [mCRPC] cohort, Mismatch Repair [MMR]/ Microsatellite Instability [MSI] defective tumours cohort and a triple negative breast cancer [TNBC] cohort) and combination expansion cohorts. In the combination expansion cohorts, TT-702 will be evaluated in combination with the androgen receptor (AR) antagonist darolutamide to be assessed in mCRPC. Potential agents for further combination expansion cohorts have not yet been defined.

The main aims of this trial are to:

* Find the maximum dose of TT-702 as a monotherapy and in combination with other anti-cancer drugs that can be given safely to patients.
* Define the side effects of TT-702 and how these can be managed.
* Determine the pharmacokinetics (PK) and elimination kinetics of TT-702.

ELIGIBILITY:
Inclusion criteria:

1. Be able to provide informed consent and be capable of co-operating with IMP administration, procedures and follow-up.
2. Be willing to provide samples (blood and tissue) as required.
3. Consent to access any available archival tissue.
4. Consent for fresh tumour biopsy samples at baseline and on trial (may be Investigator mandated for patients in the dose escalation phase; mandatory for a minimum of eight patients in each expansion cohort). Investigators will consider whether a biopsy is feasible for the patient in the dose escalation phase and this will not impede participation in the trial if biopsy is not a suitable option.
5. Life expectancy estimated by the Investigator to be at least 12 weeks.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Cohort 1M/2M (TT-702 monotherapy) - Aged 16 years or over at the time consent is given.
8. Cohort 1A/2A (TT-702 & darolutamide combination cohorts) - Aged 18 years or over at the time consent is given.
9. Haematological and biochemical indices within the protocol specified ranges.
10. Objectively or measurable evaluable disease, radiologically according to RECIST Version 1.1 (and/or, in mCRPC patients, according to PCWG3 criteria). Has radiological disease progression (and/or, in mCRPC patients, PSA progression according to PCWG3 criteria) at the time of study enrolment.
11. Castrate levels of testosterone (<1.7 nmol/L [50 ng/dL]) (mCRPC patients only).

Phase I, dose escalation phase

Histologically or cytologically proven advanced solid tumours refractory to conventional treatment, or for which no conventional therapy is considered appropriate by the Investigator or is declined by the patient. Phase I dose escalation cohorts are:

* Phase I, Cohort 1M (TT-702 monotherapy cohort): Any solid tumour for which standard of care has been exhausted or, is considered inappropriate for or, declined by the patient.
* Phase I, Cohort 1A (TT-702 & darolutamide combination cohort): mCRPC previously treated with a next generation AR antagonist (including enzalutamide, apalutamide or darolutamide) or abiraterone.
* Phase I, Cohort 1P (TT-702 & PD-1/PD-L1 combination cohort): Patients with PD-1/PD-L1 resistant tumours (i.e. disease progression after a prior PD-1/PD-L1 inhibitor with at least 12 weeks treatment).

Phase II (expansion phase)

Histologically or cytologically proven advanced solid tumour of particular interest based on preclinical and clinical data, refractory to conventional treatment or, for which no conventional therapy is considered appropriate by the Investigator or, is declined by the patient. Phase II expansion cohorts are:

• Cohort 2M (TT-702 Monotherapy expansion cohorts) - mCRPC,TNBC and MMR/MSI defective tumours:

MMR/MSI defective tumours:

* Prior treatment with an anti-PD-1 or anti-PD-L1 agent, either as monotherapy or in combination with other agent(s). This should be the preceding treatment prior to trial entry.
* Patients must have progressed on an anti-PD-1/anti-PD-L1 agent.
* Patients must have experienced Investigator-assessed initial clinical benefit from the most recent anti-PD-1/anti-PD-L1 treatment (either as monotherapy or in combination with other compounds) for at least 10 weeks. Initial benefit is defined as SD or better with an anti-PD 1/anti-PD-L1 therapy.
* Diagnosis of metastatic MSI-H (defined as MSI polymerase chain reaction test with instability shown in ≥2 or ≥30% of microsatellite markers) or metastatic MMRd (defined as loss of MLH1, MSH2, MSH6, and/or PMS2 expression is detected) through local testing in NHS lab within UKAS/ISO 15198 scope of accreditation.

mCRPC:

* Prior treatment with a next generation hormonal agent.
* Adenocarcinoma without predominant neuroendocrine or small cell features.

TNBC:

* Human epidermal growth factor receptor 2 negativity (negative immunohistochemistry [IHC] staining [score 0 or 1] or negative fluorescence in situ hybridisation based on the American Society of Clinical Oncology/College of American Pathologists guidelines and recommendations) and determined through local testing in NHS lab within UKAS/ISO 15198 scope of accreditation. Note: patients initially diagnosed with hormone receptor-positive and/ or HER2-positive breast cancer OR de novo metastatic patients with a primary tumour hormone receptor-positive (weak positivity or ER negativity and progesterone receptor positivity) considered as nonclinically relevant are eligible if the tumour biopsy obtained from a local recurrence or distant metastasis site confirms the TNBC disease.
* ER and progesterone receptor negativity (<1% positive staining cells in the invasive tumour) determined locally using IHC per American Society of Clinical Oncology/College of American Pathologists criteria.
* Patients who have received prior anti-PD-1/anti-PD-L1 agent must have experienced Investigator-assessed initial clinical benefit from the most recent anti-PD-1/anti-PD-L1 treatment (either as monotherapy or in combination with other compounds) for at least 10 weeks, followed by subsequent progression. Initial benefit is defined as SD or better with an anti-PD-1/anti-PD-L1 therapy.

Cohort 2A (TT-702 & darolutamide combination cohort): mCRPC.

* Patients with mCRPC must have progressive disease according to PCWG3 criteria.
* Previously irradiated lesions cannot be counted as target lesions unless clearly progressed after radiotherapy.
* Patients undergoing biopsy should have at least two lesions, one to be used as a target lesion and one to be biopsied.
* Cohort 2P (TT-702 & PD-1/PD-L1 combination cohort): MMR/MSI defective tumours, TNBC or mCRPC.

Exclusion criteria:

1. Radiotherapy (except single fractions for palliative reasons), endocrine therapy during the previous four weeks, immunotherapy and chemotherapy during the previous four weeks(previous six weeks for nitrosoureas, Mitomycin-C) before receiving TT-702. A washout period of eight weeks is required for enzalutamide and apalutamide before the patient receives their first dose of TT-702. A washout period of 4 weeks or 5 half-lives whichever is shorter for any other previous preceding IMPs is required before the patient receives their first dose of TT-702 (in the combination cohorts no washout is needed from PD-1/PD-L1 and darolutamide, respectively).
2. Patients with ongoing toxic manifestations of previous treatments greater than NCI CTCAE Version 5.0 Grade 1. Exceptions to this are alopecia and any ongoing toxic manifestation which in the opinion of the Investigator should not exclude the patient.
3. Patients with symptomatic brain or leptomeningeal metastases should be excluded. Asymptomatic patients with previously treated and stable brain metastases (in previous four weeks to study entry) and not requiring any steroids are eligible for the trial. Patients who are stable on anticonvulsants are also eligible.
4. Cohort 1M/2M (monotherapy) - Women of childbearing potential (or are already pregnant or lactating). However, those patients who meet the following points are considered eligible:

   • Have a negative highly sensitive pregnancy test of a serum sample within 7 days prior to trial inclusion; and

   • Agree to use two forms of medically approved contraception: i. one highly effective form including but not limited to: oral, injected,implanted, transdermal or intravaginal hormonal contraception associated with inhibition of ovulation; intrauterine device; intrauterine hormonereleasing system, bilateral tubal occlusion or vasectomised partner; ii. plus a barrier method (for example, condom plus spermicide); iii. or agree to sexual abstinence. Effective from the first administration of TT-702, throughout the trial and for six months after the last administration of IMP.
5. Male patients with partners of childbearing potential. However, those patients who meet the following points are considered eligible:

   * Agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or sexual abstinence12 effective from the first administration of IMP throughout the trial and for six months after the last administration of IMP.
   * Male patients with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicide) to prevent exposure of the foetus or neonate.
   * Non-vasectomised male patients must also be willing to ensure that any partner of childbearing potential uses a highly effective method of contraception (for example, oral, injected, implanted, transdermal or intravaginal hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system or bilateral tubal occlusion) or agree to sexual abstinence for the same duration.
6. Major thoracic or abdominal surgery from which the patient has not yet recovered.
7. At high medical risk because of non-malignant systemic disease including active uncontrolled infection. Patients with previous Hepatitis C exposure but no current infection are eligible to participate.
8. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
9. Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within eight weeks.
10. Concurrent congestive heart failure, prior history of class II-IV cardiac disease (New York Heart Association [NYHA]), prior history of clinically significant cardiac ischaemia or prior history of clinically significant cardiac arrhythmia. Patients with significant cardiovascular disease are excluded as defined by:

    1. History of congestive heart failure requiring therapy (NYHA III or IV);
    2. History of unstable angina pectoris or myocardial infarction up to six months prior to trial entry (patients with previous cardiac or thrombotic events who are now stable and or recovered are eligible);
    3. Presence of severe valvular heart disease;
    4. Presence of a ventricular arrhythmia requiring treatment;
    5. Left ventricular ejection fraction < 50%;
    6. Has a QTcF prolongation to >470 milliseconds (ms) based on a 12-lead ECG in triplicate;
    7. Previous stroke or transient ischaemic attack within 6 months of trial entry;
    8. History of clinically significant peripheral vascular disease/vasculitis/vasculopathy;
    9. Cohort 1A/2A - A history of QTcF prolongation or Torsade de pointes.
11. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I/II trial of TT-702. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP and which would not place an unacceptable burden on the patient in the opinion of the Investigator would be acceptable.
12. Previous malignancies of other types, apart from adequately treated in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for five years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
13. A concomitant significant other illness that might in the opinion of the Investigator affect compliance with the protocol or interpretation of results, examples include but are not limited to autoimmune diseases or immune deficiency, or other disease with ongoing fibrosis (such as scleroderma, pulmonary fibrosis, emphysema, neurofibromatosis, palmar/plantar fibromatosis), alcoholic hepatitis, cirrhosis, and inherited liver disease, previous organ transplantation, uncontrolled or poorly controlled diabetes mellitus (for example HbA1c >10%) and patients with non-alcoholic steatohepatitis.
14. History of an immune-mediated adverse event of Grade 3 or above attributed to prior cancer immunotherapy that resulted in permanent discontinuation of the prior immunotherapeutic agent. Immune-mediated adverse events related to prior immunomodulatory therapy (other than endocrinopathy managed with replacement therapy or stable vitiligo) that have not either resolved completely to baseline or are Grade ≤2 in severity.
15. Patients on systemic corticosteroids (apart from replacement doses for endocrinopathy up to an equivalent of 10 mg QD prednisolone). Topical or inhaled steroids for pre-existent diseases are allowed.
16. Patients who received a live vaccine within 30 days before trial enrolment are excluded.
17. Patients with a known or suspected history of hypersensitivity or allergy to TT-702, or any of its excipients (for any strength) are excluded:

    * TT-702 10 mg strength, excipients: hydroxypropyl cellulose, sodium lauryl sulfate, lactose monohydrate, microcrystalline cellulose, croscarmellose sodium and magnesium stearate;
    * TT-702 40 mg strength, excipients: hydroxypropyl cellulose, sodium lauryl sulfate, mannitol, croscarmellose sodium and magnesium stearate;
    * TT-702 120 mg strength, excipients: poloxamer-188, sodium lauryl sulfate, mannitol, croscarmellose sodium and magnesium stearate in hydroxypropyl methylcellulose (HPMC) capsules;
    * TT-478 (also known as GS-6201 or CVT-6883).
18. Cohort 1A/2A (TT-702 & darolutamide) - Patients with a known or suspected history of hypersensitivity or allergy to darolutamide or any of its excipients: calcium hydrogen phosphate, croscarmellose sodium, lactose monohydrate, magnesium stearate, povidone, hypromellose, lactose monohydrate, macrogol, and titanium dioxide.
19. Patients who take therapies that inhibit or induce CYP3A must be excluded.
20. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

If a patient is taking any dietary supplements or complementary medicines/botanicals, the Sponsor's Centre for Drug Development (CDD) must be informed at the earliest opportunity both prior to enrolment and during the patient's time on trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) (Dose Escalation Phase) | Cycle 0 Day 1 to Cycle 2 Day 1
  Determine a dose that is deemed tolerable with a target dose limiting toxicity (DLT).
Recommended Phase 2 Dose (RP2D) (Dose Escalation Phase) | Cycle 0 Day 1 to off-study visit (max. 13 months)
  The RP2D will be determined after reviewing all of the clinically relevant toxicity, efficacy and pharmacokinetic/pharmacodynamic data by the Trial Management Group.
Number of Treatment-Emergent Adverse Events (TEAEs) by Arm (Dose Escalation Phase) | Safety data will be collected from the time of informed consent until 21 days after the last dose of TT-702. The average time from consent to the end of follow up will be presented.
  Graded according to National Cancer Institute Common Criteria for Adverse Events (NCI CTCAE) Version 5.0.
Number of Grade 3, 4 and 5 TEAEs by Arm (Dose Escalation Phase) | Safety data will be collected from the time of informed consent until 21 days after the last dose of TT-702. The average time from consent to the end of follow up will be presented.
  Graded according to NCI CTCAE Version 5.0.
Number of TEAEs Related to TT-702 and/or Darolutamide by Arm (Dose Escalation Phase) | Safety data will be collected from the time of informed consent until 21 days after the last dose of TT-702. The average time from consent to the end of follow up will be presented.
  Graded according to NCI CTCAE Version 5.0.
Assess Number of Patients with Confirmed Complete Response (CR) and Partial Response (PR) (MSI/MMR and TNBC Arms Expansion Phase) | Radiological assessment within 28 days before starting TT-702; end of every 3 cycles (21-day cycles) up to 6 months then every 4 cycles & treatment discontinuation and/or off-study visit (max. 13 months)
  The number of patients who have a confirmed CR or PR according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1.
Assess Number of Patients with Confirmed CR and PR (mCRPC Arms Expansion Phase) | Radiological assessment (CT/MRI) within 28 days & bone scan (if required) within 8 weeks before starting TT-702; end of every 3 cycles (21-day cycles) up to 6 months then every 4 cycles & treatment discontinuation and/or off-study visit (max. 13 months)
  The number of patients who have a confirmed CR or PR according to Prostate Cancer Working Group 3 criteria (PCWG3) (encompassing RECIST 1.1 and Prostate Specific Antigen [PSA] level changes) in patients with mCRPC.

SECONDARY OUTCOMES:
Measurement of Maximum (or Peak) Plasma Concentration (Cmax) of TT-702 and its Active Product TT-478 as Appropriate (Dose Escalation and Expansion Phase) | From first dose of TT-702 until discontinuation visit (max. 12 months)
  Measurement of Cmax of TT-702 and its active product TT-478 as appropriate.
Measurement of Minimal Plasma Concentration (Cmin) of TT-702 and its Active Product TT-478 as Appropriate (Dose Escalation and Expansion Phase) | From first dose of TT-702 until discontinuation visit (max. 12 months)
  Measurement of Cmin of TT-702 and its active product TT-478 as appropriate.
Measurement of Time at Cmax (Tmax) of TT-702 and its Active Product TT-478 as Appropriate (Dose Escalation and Expansion Phase) | From first dose of TT-702 until discontinuation visit (max. 12 months)
  Measurement of Tmax of TT-702 and its active product TT-478 as appropriate.
Area Under the Curve (AUC) of TT-702 and its Active Product TT-478 as Appropriate (Dose Escalation and Expansion Phase) | From first dose of TT-702 until discontinuation visit (max. 12 months)
  AUC of TT-702 and its active product TT-478 as appropriate.
Apparent Clearance of TT-702 and its Active Product TT-478 as Appropriate (Dose Escalation and Expansion Phase) | From first dose of TT-702 until discontinuation visit (max. 12 months)
  Apparent clearance of TT-702 and its active product TT-478 as appropriate.
Volume of Distribution of TT-702 and its Active Product TT-478 as Appropriate (Dose Escalation and Expansion Phase) | From first dose of TT-702 until discontinuation visit (max. 12 months)
  Volume of Distribution of TT-702 and its active product TT-478 as appropriate.
Terminal Elimination Half-Life (T1/2) of TT-702 and its Active Product TT-478 as Appropriate (Dose Escalation and Expansion Phase) | From first dose of TT-702 until discontinuation visit (max. 12 months)
  T1/2 of TT-702 and its active product TT-478 as appropriate.
Assess Number of Patients with Confirmed CR and PR (Dose Escalation Phase). | Radiological assessment (CT/MRI) within 28 days & bone scan (if required) within 8 weeks before starting TT-702; end of every 3 cycles (21-day cycles) up to 6 months then every 4 cycles & treatment discontinuation and/or off-study visit (max. 13 months).
  The number of patients who have a confirmed CR or PR according to RECIST Version 1.1 or according to PCWG3 criteria (encompassing RECIST 1.1 and PSA level changes) in patients with mCRPC.
Assess Number of Patients with Confirmed CR and PR after 3, 6, 9 and 12 Cycles and at Any Time while on Trial (Dose Escalation and Expansion Phase) | Radiological assessment (CT/MRI) within 28 days & bone scan (if required) within 8 weeks before starting TT-702; end of every 3 cycles (21-day cycles) up to 6 months then every 4 cycles & treatment discontinuation and/or off-study visit (max. 13 months).
  The number of patients who have a confirmed CR or PR according to RECIST Version 1.1 or according to PCWG3 criteria (encompassing RECIST 1.1 and PSA level changes) in patients with mCRPC after 3, 6, 9 and 12 cycles and at any time while on trial.
Duration of Response and of Clinical Benefit Defined as Duration of Confirmed CR, PR or Stable Disease (SD) (Dose Escalation and Expansion Phase) | Radiological assessment (CT/MRI) within 28 days & bone scan (if required) within 8 weeks before starting TT-702; end of every 3 cycles (21-day cycles) up to 6 months then every 4 cycles & treatment discontinuation and/or off-study visit (max. 13 months).
  The duration of CR, PR or SD according to RECIST Version 1.1 or according to PCWG3 criteria (encompassing RECIST 1.1 and PSA level changes) in patients with mCRPC.
Number of Patients whose Cancer has not Progressed at Six Months (Dose Escalation and Expansion Phase ) | From first dose of TT-702 until six months after first dose of TT-702
  Number of patients whose cancer has not progressed at six months.
Number of Patients who are still Alive at 12 Months (Dose Escalation and Expansion Phase) | From first dose of TT-702 until 12 months after first dose of TT-702
  Number of patients who are still alive at 12 months.
Number of Treatment-Emergent Adverse Events (TEAEs) by Arm (Dose Expansion Phase). | Safety data will be collected from the time of informed consent until 21 days after the last dose of TT-702. The average time from consent to the end of follow up will be presented
  Graded according to NCI CTCAE version 5.0.
Number of Grade 3, 4 and 5 TEAEs by Arm (Dose Expansion Phase). | Safety data will be collected from the time of informed consent until 21 days after the last dose of TT-702. The average time from consent to the end of follow up will be presented
  Graded according to NCI CTCAE version 5.0.
Number of TEAEs Related to TT-702 and/or Darolutamide by Arm (Dose Expansion Phase) | Safety data will be collected from the time of informed consent until 21 days after the last dose of TT-702. The average time from consent to the end of follow up will be presented
  Graded according to NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, Prof, Principal Investigator — The Royal Marsden Hospital/ The Institute of Cancer Research
Locations (3):
- United Kingdom (3):
  - Royal Marsden Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitaker D, Francis L, Karaborni S, Smith S, Craigen JL, Svetlik S, Barnett S, Veal GJ. Development and validation of an LC-MS/MS method for the quantification of novel therapeutic TT-478, a selective adenosine receptor 2B antagonist, for a phase I/II clinical trial. Bioanalysis. 2025 Sep;17(17):1105-1112. doi: 10.1080/17576180.2025.2554564. Epub 2025 Oct 17. PMID 41104540